CLINICAL TRIAL: NCT02538575
Title: Prognosis Contribution of the 6 Minute Walk Test in Cystic Fibrosis : Prospective Multicenter Study
Brief Title: 6 Minute Walk Test in Cystic Fibrosis
Acronym: MUCO-TM6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Data analysis : EFFI-STAT (statistic expert) (Unknown); URC-CIC Paris Descartes Necker Cochin (Other); Funding : Association Vaincre La Mucoviscidose (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A00387-42
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Adults; 6-minute walk test
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6-minute walk test (Experimental)
  Interventions: Other: 6-minute walk test

INTERVENTIONS:
Other: 6-minute walk test — a walk of 6 minutes repeated twice in an interval of 30 minutes

SUMMARY:
The purpose of this study is to determine whether the 6-minute walk test (6MWT) could be a prognostic factor for cystic fibrosis patients.

DETAILED DESCRIPTION:
The 6-minute walk test is a simple exercise test, reproducing a daily physical activity. The utility of this test is described in several chronic lung diseases (chronic obstructive pulmonary disease, idiopathic pulmonary arterial hypertension). The distance performed during the 6MWT and / or desaturation during the 6MWT is a prognostic factor that contributes to the assessment of patients for lung transplantation indication.

The 6MWT is practiced routinely in cystic fibrosis centers but its usefulness in this disease has not been shown. Also the results of this test are not part of the decision-making criteria for lung transplantation.

A single-center study performed in adults CRCM at Cochin Hospital suggests the prognostic value of the 6MWT in patients with adult's cystic fibrosis.

The principal objective of this study is to assess the prognostic of 6MWT as part of the cystic fibrosis. The primary endpoint will be to assess the survival without lung transplant during the follow up period of 3 years. In this context, this prognostic tool could be used to help to determine the best time to consider a lung transplant in cystic fibrosis patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Cystic Fibrosis (bronchiectasis with presence of two mutations in the CFTR gene and / or positive sweat test.
* Patients aged 18 year or older.
* Pre-bronchodilator FEV1 FEV1 ≤ 60% from theoretical value: this FEV1 limits is proposed following the results from our published study (Martin et al. 2013) showing that desaturation during 6MWT and a distance ≤ 475m performed, are almost exclusively found in patients with FEV1 ≤ 60% .
* Stable health status ( >15 days after the start of treatment of a respiratory exacerbation
* No indications against the walking test:

Left uncontrolled heart failure Severe aortic stenosis acute endocarditis syncope Symptomatic severe arrhythmia stable angina Myocardial infarction <5 days Acute respiratory distress Resting SpO2≤85% pulmonary edema Uncontrolled asthma Arterial or venous thrombosis of the lower limbs, Severe acute condition that may interfere with the exercise performance (infections, renal failure, hyperthyroidism, unable to cooperate, severe pulmonary arterial hypertension, severe systemic blood pressure (Systolic blood pressure >200 mm Hg and / or diastolic blood pressure >120 mm Hg))

Exclusion Criteria:

* History of lung transplant
* Oxygen Dependence (inability to achieve a 6-minute walk test in ambient air)
* Any indication against walk test
* Pregnant women, persons deprived of liberty, person under guardianship, person in emergency situation
* Person not affiliated to social security system
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Survival without lung transplant | 3 years

SECONDARY OUTCOMES:
distance traveled during the 6MWT | one day
Oxygen desaturation (SpO2<90%) measured by a plethysmography exam during the 6MWT | one day
Number of days of intravenous antibiotic therapy | 3 years
Dyspnea questionnaire (mMRC scale) | once a year during 3 years
Measure of the Quality of life (Cystic Fibrosis Questionnaire 14+, SF12) | once a year during 3 years
Measure of Anxiety and Depression (Hospital Anxiety Depression HAD scale) | once a year during 3 years
Measure of the Physical activity (Baecke questionnaire) | once a year during 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Regis BURGEL, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, service de pneumologie, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin C, Chapron J, Hubert D, Kanaan R, Honore I, Paillasseur JL, Aubourg F, Dinh-Xuan AT, Dusser D, Fajac I, Burgel PR. Prognostic value of six minute walk test in cystic fibrosis adults. Respir Med. 2013 Dec;107(12):1881-7. doi: 10.1016/j.rmed.2013.10.001. Epub 2013 Oct 11. PMID 24157200
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Singh SJ, Puhan MA, Andrianopoulos V, Hernandes NA, Mitchell KE, Hill CJ, Lee AL, Camillo CA, Troosters T, Spruit MA, Carlin BW, Wanger J, Pepin V, Saey D, Pitta F, Kaminsky DA, McCormack MC, MacIntyre N, Culver BH, Sciurba FC, Revill SM, Delafosse V, Holland AE. An official systematic review of the European Respiratory Society/American Thoracic Society: measurement properties of field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1447-78. doi: 10.1183/09031936.00150414. Epub 2014 Oct 30. PMID 25359356